CLINICAL TRIAL: NCT00211484
Title: Treatment of Conditions With Open Label-Anecortave Acetate Sterile Suspension ( 15mg.) Where Lesions do Not Meet Acceptable Criteria for Standard Care.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA outside standard care
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Age-Related Macular Degenerations.; Subfoveal Neovascularization.
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anecortave Acetate

SUMMARY:
A compassionate method of treatment is offered to patients where lesions do not meet acceptable criteria for standard therapy. Visudyne (Photodynamic Therapy) and laser photocoagulation treatment (a treatment using heat from a fine point laser beam) have not been found to be effective in treating the lesions these patients have.

Anecortave acetate is an experimental drug that is being tested to prevent the growth of blood vessels under the retina in patients with age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Patients will receive a sub-Tenon injection of 15mg of Anecortave acetate in their study eye with the use of a counter pressure device. Patients will then be followed for up to 24 months. The patients will have the option of extending their participation in the study for an additional 24 months. Statistical analysis will include comparison of patient follow-up visual acuity and angiographic data.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of patients whose lesions do not meet acceptable criteria for standard of care treatment (PDT or laser).
2. Patients must be 18 years of age or older to receive treatment.
3. Visual acuity of 20/30 to 20/320 Study Eye on the ETDRS visual acuity chart.
4. Visual acuity of 20/800 or better Fellow Eye on the ETDRS visual acuity chart.

Exclusion Criteria:

1. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
2. Patients who have undergone intraocular surgery within last 2 months.
3. Patient participating in any other investigational drug study.
4. Use of an investigational drug or treatment related or unrelated to their condition within 30 days prior to receipt of study medication.
5. Inability to obtain photographs to document CNV (including difficulty with venous access).
6. Patient with significant liver disease or uremia.
7. Patient with known adverse reaction to fluorescein and indocyanine green or iodine.
8. Patient has a history of any medical condition which would preclude scheduled visits or completion of study.
9. Patient has had insertion of scleral buckle in the study eye.
10. Patient has received radiation treatment.
11. Patient is on anticoagulant therapy with the exception of aspirin.
12. Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2003-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
This study is designed to provide compassionate use of Anecortave Acetate Sterile Suspension of 15mg for a series of five patients where the lesions do not meet acceptable criteria for standard therapy. | 24 months

SECONDARY OUTCOMES:
mean change in VA(ETDRS), OCT, FA from baseline to 24 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason S. Slakter, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States